CLINICAL TRIAL: NCT01557543
Title: Preliminary Assessment of Direct Intra-Myocardial Injection of Autologous Bone Marrow-derived Stromal Cells on Patients Undergoing Revascularization for CAD With Depressed Left Ventricular Function
Brief Title: Stem Cell Injection to Treat Heart Damage During Open Heart Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: NIH Heart Center at Suburban Hospital (Unknown)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120078; 12-H-0078
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-06-18

CONDITIONS: Heart Disease; Ischemic Heart Disease; Coronary Artery Disease; Coronary Artery Disease (CAD)
Keywords: Coronary Artery Bypass Grafting; Coronary Artery Disease; Transmyocardial Revascularization; Bone Marrow Stromal Cells
MeSH Terms: conditions — Heart Diseases; Myocardial Ischemia; Coronary Artery Disease | interventions — Cell- and Tissue-Based Therapy

INTERVENTIONS:
Other: Cell Therapy — Intramyocardial Injection of BMSCs

SUMMARY:
Background:

- Bone marrow stromal stem cells (also known as mesenchymal stem cells) have been isolated and are found to make large amounts of growth factors. Because they make growth factors, these cells can help re-grow tissue and encourage repair of damaged tissue. Tests on damaged heart muscle suggest that injecting these cells directly into damaged heart muscle can improve heart function. Researchers want to give stem cells to people who are having open heart surgery to see if they can help to repair heart muscle damage.

Objectives:

- To test the safety and effectiveness of bone marrow stromal stem cell injections given during heart surgery to treat heart muscle damage.

Eligibility:

- Individuals at least 18 years of age who are scheduled to have open heart surgery for heart artery or vein blockages.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will also be collected.
* Participants will have bone marrow taken from both hip bones about 3 weeks before the heart surgery.
* During the surgery, the stromal stem cells collected from the bone marrow will be given into the damaged portion of the heart muscle. The rest of the heart surgery will be performed according to standard procedures.
* After the surgery, participants will be monitored for complications from the stromal stem cells.
* Participants will have heart function tests to see if the stromal stem cell treatments were effective....

DETAILED DESCRIPTION:
Background:

Many investigators now believe that bone marrow-derived stem cells or endothelial progenitor cells can be recruited to and incorporated into tissues undergoing neovascularization, including cardiac tissue.

Stem cells which include hematopoietic stem cells (HSCs), endothelial progenitor cells (EPCs), mesenchymal stem cells / stromal stem cells (MSCs), myoblasts, and undifferentiated side population cells have been used as an alternative therapeutic strategy for ischemic cardiovascular diseases that cannot be treated by routine interventional approaches.

In a porcine pre-clinical study we found that cells survived after intramyocardial injection and differentiated into vascular cells, smooth muscle or endothelial cells. Functional analysis of regional wall motion and ejection fraction demonstrated statistically significant improvement in function in cell treated animals after six weeks compared with baseline and sham controls.

A variety of studies have been conducted in subjects with coronary artery disease using different cell types and routes of administration. This study will be the first of its kind to administer autologous BMSC via direct intramyocardial injection in a rigorous clinical trial in the U.S.

Objectives:

To evaluate the safety and feasibility of direct intra-myocardial injection of autologous bone marrow stromal cells (BMSCs) in adult subjects undergoing coronary artery bypass graft (CABG) or transmyocardial revascularization (TMR).

A secondary objective is to assess whether direct intra-myocardial injection of autologous bone marrow stromal cells (BMSCs) improves the patient s cardiac function, quality of life, and reduces cardiac events compared with historical controls at three and six months after intervention.

Eligibility:

Adult subjects with three-vessel coronary artery disease who plan to undergo CABG or TMR at the NIH Heart Center at Suburban Hospital and are willing to participate, who have stable angina, LV EF less than or equal to 50%, and who have evidence of hypokinetic segments.

Subjects will be excluded if they have had a recent myocardial infarction (MI), bleeding disorder, infection, HIV or who are unable to wait 3 weeks for surgery while cells are being expanded prior to injection.

Design:

Bone marrow aspiration will be performed on subjects who suffer from ischemic heart disease with depressed left ventricular function three weeks before their admission to have CABG or TMR in the NIH Clinical Center Outpatient Clinic.

Data will be presented based on the subject s treatment regimen:

Group 1 CABG+Cells (total of 10 evaluable subjects)

Group 2 TMR + Cells (total of 10 evaluable subjects)

The autologous MSCs will be isolated from the marrow aspirate, cultured and expanded in vitro for 3 passages (approximately 21 days (+/- 4 days)) in the Clinical Center Cell Processing Laboratory (CPS), located in the Department of Transfusion Medicine (DTM), Clinical Center, NIH.

During the surgery at Suburban Hospital, the MSCs will be injected directly into the ischemic area after CABG or TMR. Patients will be assessed for functional improvements pre, 3, 6, 12 and 60 months after the surgery by transthoracic echocardiography and/or by MRI at pre, 3 and 6 months after surgery. Toxicity data will be reported from time of surgery to 6 months after surgery, unless later toxicities occur that are related to cell injection.

ELIGIBILITY:
* INCLUSION CRITERIA
* Consenting adult patients (male or female, aged above 18 and less than or equal to 85), and
* Plans to undergo CABG or TMR at the NIH Heart Center at Suburban Hospital and are willing to participate.
* Must meet indications for CABG or TMR:
* Indications for CABG (31)

  1. Significant left main coronary artery stenosis (> 50% reduction in lumen diameter).
  2. Left main equivalent: significant (greater than or equal to70%) stenosis of proximal LAD and proximal left circumflex artery.
  3. Three-vessel disease (stenosis of 50% or more in all 3 major coronary territories). (Survival benefit is greater when LVEF is

     <0.50.)
  4. Two-vessel disease with significant proximal LAD stenosis and either EF <0.50 or demonstrable ischemia on noninvasive

     testing.
  5. One- or 2-vessel coronary artery disease without significant proximal LAD stenosis, but with a large area of viable

myocardium and high-risk criteria on noninvasive testing.

- Indications for TMR (32, 33).

1. Canadian Cardiovascular Class III or IV angina that is refractory to maximal medical therapy.
2. Reversible ischemia of the left ventricular free wall and coronary artery disease corresponding to the regions of myocardial

   ischemia.
3. In all regions of the myocardium, the coronary disease must not be amenable to coronary artery bypass graft (CABG) or

percutaneous transluminal coronary angioplasty (PTCA), due to:

i. severe diffuse disease,

ii. lack of suitable targets for complete revascularization,

iii. lack of suitable conduits for complete revascularization

- Stable Angina. Patient?s clinical state has to be stable to receive surgical treatment. Patients must have received or currently receiving standard of care medical therapy(33) for at least 4 weeks prior to enrollment, to include:

1. Aspirin in the absence of contraindications in patients with prior MI
2. Beta-blockers as initial therapy in the absence of contraindications in patients with prior MI.
3. Lipid-lowering therapy in patients with documented CAD and LDL cholesterol greater than 130 mg/dL, with a target LDL of less

   than 100 mg/dL
4. ACE inhibitor in patients with CAD (considered significant by angiography or previous MI) who also have diabetes and/or left

ventricular systolic dysfunction.

* Three-vessel CAD. Multi-vessel diffuse coronary artery disease not amenable to percutaneous coronary intervention.
* LV EF less than or equal to 50% by by MRI or Echocardiogram. The left ventricle ejection fraction less than 50% evidenced the diagnosis of heart failure indicating global weakness of myocardial contractility and leaves space for functional improvement.
* Evidence of hypokinetic segment. Regional wall motion abnormality which includes regional low/no motion, or motion in opposite direction, is a good indication for invasive intervention and can be well-compared before and after treatment.
* Laboratory tests showed no evidence of major organ dysfunction, bleeding disorder, or infectious diseases. Patients must have organ and marrow function as defined below:

  i. Leukocytes greater than or equal to 2,500/mcL

ii. Lymphocytes greater than or equal to 800/mcL

iii. Platelets greater than or equal to 100,000/mcL

iv. Total Bilirubin less than or equal to 2mg/dL

v. AST (SGOT)/ALT (SGPT) less than or equal 1.5 times

institutional upper limit of normal (ULN)

vi. Creatinine less than or equal to institutional upper limit of

normal (ULN)

* Must be willing to participate in 10-CC-0053 to obtain autologous bone marrow.
* Patients must understand and sign an informed consent document that explains the nature of his/her cardiac disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, and potential risks and toxicities.

EXCLUSION CRITERIA

* Patients who have the following conditions will be excluded from the study:
* Acute MI. Less than three months after recent acute myocardial infarction.
* Unstable angina. Excluded due to the propensity to deteriorate into AMI.
* Bleeding disorder, including history of familial hemophilia, signs and symptoms of easy bruising, petechiae, or platelet count < 80,000 cells/mcL. This disorder may unnecessarily complicate the operative procedure and postoperative recovery.
* Severe respiratory disorder, including acute asthma, chronic bronchitis, severe chronic obstructive lung disease. A disorder that would complicate the operative procedure and postoperative recovery.
* Unable to provide informed consent on this study or on 10-CC-0053.
* Unable to wait 3 weeks for surgery, which is the waiting period for ex-vivo cell expansion.
* Reactive for anti-HIV, Hepatitis B surface antigen, anti-HCV or nucleic acid testing for HIV, Hepatitis B and C. An investigational component accompanying this major surgical procedure in the presence of infection has the potential to increase risk of complications, and manufacturing contaminated products risks contaminating other cellular products in CPS.
* Pregnant or lactating females, due to the highly investigational nature of this study and its unknown effects on a developing fetus.
* Allergic to Gentamicin.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02-29; Primary Completion 2017-07-25 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and feasibility of direct intra-myocardial injection of autologous bone marrow stromal cells (BMSCs) in adult subjects undergoing coronary artery bypass graft (CABG) or transmyocardial revascularization (TMR).

SECONDARY OUTCOMES:
To assess if direct intra-myocardial injection of autologous BMSCs improves the patient's cardiac function, quality of life, and reduces cardiac events compared to historical controls at three and six months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela G Robey, Ph.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Suri C, Jones PF, Patan S, Bartunkova S, Maisonpierre PC, Davis S, Sato TN, Yancopoulos GD. Requisite role of angiopoietin-1, a ligand for the TIE2 receptor, during embryonic angiogenesis. Cell. 1996 Dec 27;87(7):1171-80. doi: 10.1016/s0092-8674(00)81813-9. PMID 8980224
- [Background] Assmus B, Schachinger V, Teupe C, Britten M, Lehmann R, Dobert N, Grunwald F, Aicher A, Urbich C, Martin H, Hoelzer D, Dimmeler S, Zeiher AM. Transplantation of Progenitor Cells and Regeneration Enhancement in Acute Myocardial Infarction (TOPCARE-AMI). Circulation. 2002 Dec 10;106(24):3009-17. doi: 10.1161/01.cir.0000043246.74879.cd. PMID 12473544
- [Background] Britten MB, Abolmaali ND, Assmus B, Lehmann R, Honold J, Schmitt J, Vogl TJ, Martin H, Schachinger V, Dimmeler S, Zeiher AM. Infarct remodeling after intracoronary progenitor cell treatment in patients with acute myocardial infarction (TOPCARE-AMI): mechanistic insights from serial contrast-enhanced magnetic resonance imaging. Circulation. 2003 Nov 4;108(18):2212-8. doi: 10.1161/01.CIR.0000095788.78169.AF. Epub 2003 Oct 13. PMID 14557356